CLINICAL TRIAL: NCT06228417
Title: Adaptive Digital Interventions Through Mobile App for Medication Adherence Improvement in Persons With Hypertension: a Pilot Study for Usability
Brief Title: A Mobile App for Medication Adherence in Persons With Hypertension: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Halmstad University (Other)
Collaborators: Vinnova (Other Government)
Responsible Party: Principal Investigator, Slawomir Nowaczyk, Professor, Halmstad University
Other Study IDs: 2017_04617
Record Dates: First submitted 2023-12-27; First posted 2024-01-29 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
Keywords: artificial intelligence; focus group; adherence, medication; pilot study
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adaptive digital intervention — Participants received reminder for medication intake on daily basis. Also, short message regarding hypertension, medication and lifestyle changes

SUMMARY:
A development and pilot test of an app targeting persons with hypertension. Content in the app was based on persons with hypertensions experiences and a literature review. The participants experience of using the app as well as testing a instrument for medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* 40-70 years of age,
* have hypertension (i.e., ICD 10 codes I10-I15 in the person's medical history) for ≥1 year
* have been prescribed medications to treat said hypertension
* speak and understand Swedish
* have a smartphone

Exclusion Criteria:

* having received medication with unit-dose packages (Apodos)
* previous stroke
* previous myocardial infarction
* psychological disorder or cognitive impairment (i.e. ICD 10 codes F01-F99)
* pregnancy-induced hypertension´
* insulin treatment
* kidney disease, defined as glomerulus filtration rate (GFR) <60 ml/min.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with hypertension, more than one year, were enrolled. From primary care.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-02-23 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence | two weeks
  Medication adherence measured by the participants self-reported intake of daily medication in the app.
  The usage is described in frequencies and response time.
Adherence hypertension medication | two weeks
  Medication score through the Maastricht Utrecht Adherence in Hypertension (MUAH-16) questionnaire.
  The questionnaire consists of four subscales: two of them measures positive and two others measures negative aspects of attitudes to medication adherence and health problem. Min value for each subscale are 4 and maximum 28. Higher value indicate better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Nowaczyk, Professor, Principal Investigator — Halmstad University
Locations (1):
- Halmstad University, Halmstad, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Only researchers included in the study the will have access.